CLINICAL TRIAL: NCT02793050
Title: Trabectedin in Soft Tissue Sarcomas. A Retrospective Observational Analysis (TrObs)
Brief Title: Retrospective Study of Trabectedin in Soft Tissue Sarcomas
Acronym: TrObs
Status: Completed | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ISG TrObs
Record Dates: First submitted 2016-05-25; First posted 2016-06-08 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Trabectedin; Soft Tissue Sarcoma; Observational
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trabectedin: Trabectedin give according the market authorization for advanced soft tissue sarcoma
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Collection of data on the clinical use of Trabectedin
  Other Names: yondelis

SUMMARY:
This is an independent, observational, retrospective post marketing study on the use of trabectedin in a clinical setting.

A data collection on the clinical use of the drug will help to improve knowledge and might contribute to optimize the clinical use of the drug.

DETAILED DESCRIPTION:
This is a national, multi-centre observational retrospective and prospective chart review study of treatment patterns and clinical outcomes in a subset of patients with Soft Tissue Sarcoma who received trabectedin as per licensed indication.

In the absence of availability of existing databases, a retrospective chart review design was selected.

It is anticipated that the medical charts will contain the information required to answer study objectives. This chart review study will be conducted in 25 sites in Italy An estimated total of 900 charts will be abstracted. This study requires no intervention or interference with standard medical care, and thus it will not affect patient treatment.

The study is sponsored by Italian Sarcoma Group Charts of patients who initiated trabectedin as part of the approved treatment for a Soft Tissue Sarcoma , will be identified by site staff. Each identified chart will be assigned a unique study identification number. Site staff will review the medical charts for all identified patients to determine patient eligibility. Those patients who meet eligibility criteria will be enrolled into the final study cohort as subject.

Data from subject medical charts will be abstracted by local site study staff and entered at the site into an electronic data capture (EDC) system. The system will also facilitate the monitoring of the completeness and quality of study data as the study data accrue.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received trabectedin according to the approved indication in the period January 2010 December 2015

Exclusion Criteria:

* Trabectedin started before January 2010 and after December 2015
* Participation into clinical trials with trabectedin
* Clinical chart missing, empty, or not retrievable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced soft tissue sarcoma who received trabectedin according its market authorisation, in Italy from 01Jan2010 to 31Dec2015
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Post-trabectedin received treatment | Through treatment completion, an average of 24 month
  Number of chemotherapy lines received after trabectedin given according to the approved indication

SECONDARY OUTCOMES:
Tumor response | after 6 months from trabectedin start date
  Percent of patients with non progressing disease at 6 months
Trabectedin dose modification | Through treatment completion, an average of 24 month
  Describe trabectedin treatment experience in term of dose for patients with Soft Tissue Sarcoma treated with trabectedin as per market indication
Progression-free survival | after 5 years and 3 years from trabectedin start date
  Describe progression-free survival (PFS) for patients with Soft Tissue Sarcoma who received trabectedin.
Trabectedin safety profile | Through treatment completion, an average of 24 month
  Describe trabectedin safety profile in terms of number of participants with treatment-related adverse events as assessed by CTCAE v4.0 tha caused treatment discontinuation
Overall survival | after 5 years and 3 years from trabectedin start date
  Describe overall survival (OS) for patients with Soft Tissue Sarcoma who received trabectedin.

OTHER OUTCOMES:
Histology related treatment response | after 6 months from trabectedin start date
  Number of patient who did not progress based on the different Soft Tissue Sarcoma histology sub-type

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ferrari, MD, Principal Investigator — Italian Sarcoma Group
Locations (26):
- Italy (26):
  - A.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Istituto Tumori Giovanni Paolo II, Bari, BA
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Ospedale Oncologico A. Businco, Cagliari, CA
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola, FC
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Centro di Riferimento Oncologico di Aviano, Aviano, PD
  - Istituto Oncologico Veneto, Padua, PD
  - Azienda Ospedaliera Universitaria Santa Chiara, Pisa, PI
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Istituto Ortopedico Rizzoli, Bologna
  - Policlinico S.Orsola Malpighi - Unit of Medical Oncology, Bologna
  - Pres.Ospedal.Spedali Civili Brescia -, Brescia (BS)
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Irccs Istituto Nazionale Dei Tumori (Int), Milano (MI)
  - Azienda Ospedaliero-Universitaria di Modena - Policlinico, Modena
  - Irccs Istituto Nazionale Tumori Fondazione Pascale -, Napoli (NA)
  - Ospedale Misericordia e Dolce Ist. Toscano Tumori, Az. USL4, Prato
  - Arcispedale S. Maria Nuova Azienda Ospedaliera Di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario "Agostino Gemelli", Roma
  - Istituto Regina Elena - IFO, Rome
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - Presidio Sanitario Gradenigo Di Torino, Torino (TO)

IPD SHARING:
Plan to Share IPD: Yes
Aggregate anonymized results will be available upon request at the end of the study

REFERENCES:
- [Background] Stiller CA, Trama A, Brewster DH, Verne J, Bouchardy C, Navarro C, Chirlaque MD, Marcos-Gragera R, Visser O, Serraino D, Weiderpass E, Dei Tos AP, Ascoli V; RARECARE Working Group. Descriptive epidemiology of Kaposi sarcoma in Europe. Report from the RARECARE project. Cancer Epidemiol. 2014 Dec;38(6):670-8. doi: 10.1016/j.canep.2014.09.009. Epub 2014 Oct 22. PMID 25454979
- [Background] ESMO/European Sarcoma Network Working Group. Soft tissue and visceral sarcomas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2014 Sep;25 Suppl 3:iii102-12. doi: 10.1093/annonc/mdu254. No abstract available. PMID 25210080
- [Background] Judson I, Verweij J, Gelderblom H, Hartmann JT, Schoffski P, Blay JY, Kerst JM, Sufliarsky J, Whelan J, Hohenberger P, Krarup-Hansen A, Alcindor T, Marreaud S, Litiere S, Hermans C, Fisher C, Hogendoorn PC, dei Tos AP, van der Graaf WT; European Organisation and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Doxorubicin alone versus intensified doxorubicin plus ifosfamide for first-line treatment of advanced or metastatic soft-tissue sarcoma: a randomised controlled phase 3 trial. Lancet Oncol. 2014 Apr;15(4):415-23. doi: 10.1016/S1470-2045(14)70063-4. Epub 2014 Mar 5. PMID 24618336
- [Background] Sleijfer S, Ouali M, van Glabbeke M, Krarup-Hansen A, Rodenhuis S, Le Cesne A, Hogendoorn PC, Verweij J, Blay JY. Prognostic and predictive factors for outcome to first-line ifosfamide-containing chemotherapy for adult patients with advanced soft tissue sarcomas: an exploratory, retrospective analysis on large series from the European Organization for Research and Treatment of Cancer-Soft Tissue and Bone Sarcoma Group (EORTC-STBSG). Eur J Cancer. 2010 Jan;46(1):72-83. doi: 10.1016/j.ejca.2009.09.022. PMID 19853437
- [Background] Italiano A, Mathoulin-Pelissier S, Cesne AL, Terrier P, Bonvalot S, Collin F, Michels JJ, Blay JY, Coindre JM, Bui B. Trends in survival for patients with metastatic soft-tissue sarcoma. Cancer. 2011 Mar 1;117(5):1049-54. doi: 10.1002/cncr.25538. Epub 2010 Oct 13. PMID 20945333
- [Background] Pommier Y, Kohlhagen G, Bailly C, Waring M, Mazumder A, Kohn KW. DNA sequence- and structure-selective alkylation of guanine N2 in the DNA minor groove by ecteinascidin 743, a potent antitumor compound from the Caribbean tunicate Ecteinascidia turbinata. Biochemistry. 1996 Oct 15;35(41):13303-9. doi: 10.1021/bi960306b. PMID 8873596
- [Background] Bonfanti M, La Valle E, Fernandez Sousa Faro JM, Faircloth G, Caretti G, Mantovani R, D'Incalci M. Effect of ecteinascidin-743 on the interaction between DNA binding proteins and DNA. Anticancer Drug Des. 1999 Jun;14(3):179-86. PMID 10500494
- [Background] Erba E, Bergamaschi D, Bassano L, Damia G, Ronzoni S, Faircloth GT, D'Incalci M. Ecteinascidin-743 (ET-743), a natural marine compound, with a unique mechanism of action. Eur J Cancer. 2001 Jan;37(1):97-105. doi: 10.1016/s0959-8049(00)00357-9. PMID 11165136
- [Background] Fayette J, Coquard IR, Alberti L, Boyle H, Meeus P, Decouvelaere AV, Thiesse P, Sunyach MP, Ranchere D, Blay JY. ET-743: a novel agent with activity in soft-tissue sarcomas. Curr Opin Oncol. 2006 Jul;18(4):347-53. doi: 10.1097/01.cco.0000228740.70379.3f. PMID 16721129
- [Background] D'Incalci M, Badri N, Galmarini CM, Allavena P. Trabectedin, a drug acting on both cancer cells and the tumour microenvironment. Br J Cancer. 2014 Aug 12;111(4):646-50. doi: 10.1038/bjc.2014.149. Epub 2014 Apr 22. PMID 24755886
- [Background] Garcia-Carbonero R, Supko JG, Maki RG, Manola J, Ryan DP, Harmon D, Puchalski TA, Goss G, Seiden MV, Waxman A, Quigley MT, Lopez T, Sancho MA, Jimeno J, Guzman C, Demetri GD. Ecteinascidin-743 (ET-743) for chemotherapy-naive patients with advanced soft tissue sarcomas: multicenter phase II and pharmacokinetic study. J Clin Oncol. 2005 Aug 20;23(24):5484-92. doi: 10.1200/JCO.2005.05.028. PMID 16110008
- [Background] Garcia-Carbonero R, Supko JG, Manola J, Seiden MV, Harmon D, Ryan DP, Quigley MT, Merriam P, Canniff J, Goss G, Matulonis U, Maki RG, Lopez T, Puchalski TA, Sancho MA, Gomez J, Guzman C, Jimeno J, Demetri GD. Phase II and pharmacokinetic study of ecteinascidin 743 in patients with progressive sarcomas of soft tissues refractory to chemotherapy. J Clin Oncol. 2004 Apr 15;22(8):1480-90. doi: 10.1200/JCO.2004.02.098. PMID 15084621
- [Background] Le Cesne A, Ray-Coquard I, Duffaud F, Chevreau C, Penel N, Bui Nguyen B, Piperno-Neumann S, Delcambre C, Rios M, Chaigneau L, Le Maignan C, Guillemet C, Bertucci F, Bompas E, Linassier C, Olivier T, Kurtz JE, Even C, Cousin P, Yves Blay J; French Sarcoma Group. Trabectedin in patients with advanced soft tissue sarcoma: a retrospective national analysis of the French Sarcoma Group. Eur J Cancer. 2015 Apr;51(6):742-50. doi: 10.1016/j.ejca.2015.01.006. Epub 2015 Feb 23. PMID 25727882
- [Background] Demetri GD, Chawla SP, von Mehren M, Ritch P, Baker LH, Blay JY, Hande KR, Keohan ML, Samuels BL, Schuetze S, Lebedinsky C, Elsayed YA, Izquierdo MA, Gomez J, Park YC, Le Cesne A. Efficacy and safety of trabectedin in patients with advanced or metastatic liposarcoma or leiomyosarcoma after failure of prior anthracyclines and ifosfamide: results of a randomized phase II study of two different schedules. J Clin Oncol. 2009 Sep 1;27(25):4188-96. doi: 10.1200/JCO.2008.21.0088. Epub 2009 Aug 3. PMID 19652065
- [Background] Grosso F, Sanfilippo R, Virdis E, Piovesan C, Collini P, Dileo P, Morosi C, Tercero JC, Jimeno J, D'Incalci M, Gronchi A, Pilotti S, Casali PG. Trabectedin in myxoid liposarcomas (MLS): a long-term analysis of a single-institution series. Ann Oncol. 2009 Aug;20(8):1439-44. doi: 10.1093/annonc/mdp004. Epub 2009 May 22. PMID 19465423
- [Background] Samuels BL, Chawla S, Patel S, von Mehren M, Hamm J, Kaiser PE, Schuetze S, Li J, Aymes A, Demetri GD. Clinical outcomes and safety with trabectedin therapy in patients with advanced soft tissue sarcomas following failure of prior chemotherapy: results of a worldwide expanded access program study. Ann Oncol. 2013 Jun;24(6):1703-9. doi: 10.1093/annonc/mds659. Epub 2013 Feb 5. PMID 23385197
- [Background] Blay JY, Italiano A, Ray-Coquard I, Le Cesne A, Duffaud F, Rios M, Collard O, Bertucci F, Bompas E, Isambert N, Chaigneau L, Cassier P, Bui B, Decanter G, Derbel O, Coindre JM, Zintl P, Badri N, Penel N. Long-term outcome and effect of maintenance therapy in patients with advanced sarcoma treated with trabectedin: an analysis of 181 patients of the French ATU compassionate use program. BMC Cancer. 2013 Feb 6;13:64. doi: 10.1186/1471-2407-13-64. PMID 23388156
- [Background] Le Cesne A, Blay JY, Domont J, Tresch-Bruneel E, Chevreau C, Bertucci F, Delcambre C, Saada-Bouzid E, Piperno-Neumann S, Bay JO, Mir O, Ray-Coquard I, Ryckewaert T, Valentin T, Isambert N, Italiano A, Clisant S, Penel N. Interruption versus continuation of trabectedin in patients with soft-tissue sarcoma (T-DIS): a randomised phase 2 trial. Lancet Oncol. 2015 Mar;16(3):312-9. doi: 10.1016/S1470-2045(15)70031-8. Epub 2015 Feb 11. PMID 25680558
- [Derived] Palmerini E, Sanfilippo R, Grignani G, Buonadonna A, Romanini A, Badalamenti G, Ferraresi V, Vincenzi B, Comandone A, Pizzolorusso A, Brunello A, Gelsomino F, De Pas T, Ibrahim T, Gurrieri L, Grosso F, Zanelli F, Pantaleo MA, Milesi L, Ciuffreda L, Ferrari V, Marchesi E, Quattrini I, Righi A, Setola E, Carretta E, Casali PG, Picci P, Ferrari S. Transcription regulators and ultra-rare and other rare translocation-related sarcomas treated with trabectedin: A proof of principle from a post-hoc analysis. Front Oncol. 2022 Dec 8;12:1042479. doi: 10.3389/fonc.2022.1042479. eCollection 2022. PMID 36568164
- [Derived] Palmerini E, Sanfilippo R, Grignani G, Buonadonna A, Romanini A, Badalamenti G, Ferraresi V, Vincenzi B, Comandone A, Pizzolorusso A, Brunello A, Gelsomino F, Pas T, Ibrahim T, Grosso F, Zanelli F, Pantaleo MA, Milesi L, Ciuffreda L, Ferrari V, Marchesi E, Quattrini I, Righi A, Setola E, Carretta E, Picci P, Ferrari S. Trabectedin for Patients with Advanced Soft Tissue Sarcoma: A Non-Interventional, Retrospective, Multicenter Study of the Italian Sarcoma Group. Cancers (Basel). 2021 Mar 2;13(5):1053. doi: 10.3390/cancers13051053. PMID 33801399